CLINICAL TRIAL: NCT03683420
Title: Using Music As a Tool for Distress Reduction During Cancer Treatment
Brief Title: Music in Reducing Distress in Participants with Cancer During Chemotherapy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Felicity Harper, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-130; NCI-2018-00454 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-130 (Other: Wayne State University/Karmanos Cancer Institute)
Record Dates: First submitted 2018-04-22; First posted 2018-09-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Caregiver; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (music) (Experimental): The intervention is a behavioral intervention, which consists of giving patients and caregivers iPods to listen to music for up to 60 minutes while the patient is receiving a chemo infusion. The study consists of a presurvey, active listening period, and a post-survey.
  Interventions: Behavioral: Music Therapy
- Group II (control) (No Intervention): The intervention is a behavioral intervention, which consists of giving patients and caregivers iPods to listen to music for up to 60 minutes while the patient is receiving a chemo infusion. Participants and caregivers in the control condition complete a presurvey and post survey but do not listen to music during infusion session .

INTERVENTIONS:
Behavioral: Music Therapy — The intervention consists of using an iPod to listen to music for up to 60 minutes while patients are receiving chemo infusion. There are no on components to the study.
  Arms: Group I (music)

SUMMARY:
This trial studies how well music works in reducing distress in participants with cancer during chemotherapy treatment. Music in participants receiving cancer treatment such as infusion treatment and caregiver may reduce pain, anxiety, and distress and improve participant's psychological and physiological wellbeing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the effect of patients? listening to music on level of distress during cancer treatment.

SECONDARY OBJECTIVES:

I. To explore the influence of covariates (patients? sociodemographics, musical background, and clinical variables) on the association between patients? listening to music and level of distress during cancer treatment.

II. To explore the interdependence of adjustment among patients and their caregivers on the association between.

OUTLINE: Participants and caregivers are randomized to 1 of 2 groups.

GROUP I: Participants and caregivers listen to music of their choice for up to 60 minutes during infusion session.

GROUP II: Participants and caregivers do not listen to music during infusion session and are placed on music waitlist.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, write and understand English
* Have sufficient hearing capacity to hear music

Exclusion Criteria:

* Patients with cognitive or perceptual disturbances will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in pain assessed by Visual Analogue Scale | 1 hour
  Clinical variables will be summarized by median and range for continuous variables and by count and percentage for categorical variables. The changes between pre- and post-survey will be compared between control and experimental groups using an unpaired t-test. Total scores are reported with the total scores ranging from 0-10; higher scores indicate more pain.
Changes in mood assessed by Positive and Negative Affect Scale | 1 hour
  Clinical variables will be summarized by median and range for continuous variables and by count and percentage for categorical variables. The changes between pre- and post-survey will be compared between control and experimental groups using an unpaired t-test. There are two subscales: Positive Affect and Negative Affect. Scores for each subscale (10 items each) range from 10 to 50 with higher scores meaning higher levels of affect (either higher positive or higher negative affect).
Changes in distress assessed by Distress Thermometer. | 1 hour
  Clinical variables will be summarized by median and range for continuous variables and by count and percentage for categorical variables. The changes between pre- and post-survey will be compared between control and experimental groups using an unpaired t-test. Total scores are reported with the total scores ranging from 0-10; higher scores indicate more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Felicity Harper, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Harper FWK, Heath AS, Moore TF, Kim S, Heath EI. Using Music as a Tool for Distress Reduction During Cancer Chemotherapy Treatment. JCO Oncol Pract. 2023 Dec;19(12):1133-1142. doi: 10.1200/OP.22.00814. Epub 2023 Jul 11. PMID 37433094